CLINICAL TRIAL: NCT05755373
Title: A Multinational Survey-based Study to Understand the Real-world Awareness and Perceptions of Systemic inFLAMmation and rolE of hsCRP as a Biomarker in Patients With AtheroSclerotic CardioVascular Disease and Chronic Kidney Disease Among Cardiologists
Acronym: FLAME-ASCVD
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7672; U1111-1284-5885 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD); Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Atherosclerosis; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiologists: Cardiologists treating patients with ASCVD and CKD
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The purpose of this survey is to collect information for scientific research and to better understand the role of systemic inflammation in identification, treatment and management of patients with ASCVD and CKD.

This study is a cross-sectional design conducted among cardiologists in United Kingdom, Italy, Germany, Brazil, Saudi Arabia, Japan, Australia, China, India and France, treating ASCVD and CKD patients. Study participants will be recruited to complete an approximately 20-minute self-administered online survey. Recruitment will be conducted through email and phone. Data is collected though online data collection using a programmed survey.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age above or equal to 18 years at the time of signing informed consent.
3. Is a Cardiologist.
4. Has been in practice greater than or equal to 3 years.
5. Sees at least 15 ASCVD and CKD patients per month.

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
3. Does not meet inclusion criteria requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiologists treating patients with ASCVD and CKD
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Cardiologists' perceptions towards the role of systemic inflammation in the identification, treatment and management of patients with ASCVD and CKD. Multi-select from a defined list. | At the time of survey response (Day 1)
  Numerical; A 7-point Likert scale for measurement of agreement from 1 "strongly disagree" to 7 "strongly agree".

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bangalore, India

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com